CLINICAL TRIAL: NCT01943578
Title: Prospective Observational Cohort Study of the Value of the Six Minute Walk Test and Handgrip Strength in Lung Cancer Patients Undergoing Chemotherapy
Brief Title: Value of Physical Capacity Tests in Lung Cancer
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Morten Quist, phd student, Rigshospitalet, Denmark
Other Study IDs: 2007-58-0015-30-1059
Record Dates: First submitted 2013-08-30; First posted 2013-09-17 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Non Small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lung cancer patients: Non Small Cell Lung Cancer, Small Cell Lung Cancer

SUMMARY:
The study examines the physical capacity of lung cancer patients assessed with the six minute walk test and handgrip strength. Demographic and selfreported exercise behavior is registered to explore correlations to functional and physical capacity.

Assessments are made before first chemotherapy cycle and after fourth chemotherapy cycle, an expected average of 12 weeks between first and second assessment.

ELIGIBILITY:
Inclusion Criteria:

* Non small cell lung cancer stage I-IV
* Small cell lung cancer
* Patients >18 years
* WHO performance status 0-2
* undergoing chemotherapy

Exclusion Criteria:

* unstable angina during the previous month
* myocardial infarction diagnosed within the last month
* not approval for physical activity by primary oncologist
* inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non Small Cell Lung Cancer Stage Small Cell Lung Cancer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mortality - Survival time | time from first chemotherapy treatment to death, assessed after 30 months
  Prognostic value of the six minute walk and handgrip strength on mortality

SECONDARY OUTCOMES:
Hand grip strength | before first chemotherapy and after fourth cycle of chemotherapy, an expected average of 12 weeks between first and second assessment.
Self reported exercise behavior | before first chemotherapy and after fourth cycle of chemotherapy, an expected average of 12 weeks between first and second assessment.
Six minute walk test | Before first and after fourth chemotheraphy cycle, an expected average of 12 weeks between first and second assessment.

OTHER OUTCOMES:
FACT-L | Before first chemotherapy and after fourth cycle of chemotherapy, an expected average of 12 weeks between first and second assessment.
  Patient reported outcome

CONTACTS AND LOCATIONS:
Overall Officials: Seppo Langer, Phd., Study Chair — University Hospital of Copenhagen, Rigshospitalet
Locations (1):
- University Hospital of Copenhagen, Copenhagen, Denmark

REFERENCES:
- See also: Related Info — http://www.ucsf.dk/